CLINICAL TRIAL: NCT01424488
Title: Randomized, Parallel-group, Placebo-controlled, Safety-assessor Blinded Trial in Adult Subjects Evaluating the Efficacy and Safety of Sugammadex for Reversal of Pipecuronium-induced Neuromuscular Blockade in Subjects Undergoing Abdominal Surgery Under General Anesthesia
Brief Title: Sugammadex Efficacy and Safety for Reversal of Pipecuronium-induced Neuromuscular Blockade
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Clinical Hospital #1 of LLC Russian Railways (Other Government)
Responsible Party: Principal Investigator, Eduard Nikolaenko, Professor Nikolaenko, Central Clinical Hospital #1 of LLC Russian Railways
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCHRussianRailways
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Adult Subjects Undergoing Abdominal Surgery Under General Anesthesia
Keywords: sugammadex; reversal; pipecuronium-induced neuromuscular blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugammadex group (Experimental): 4 mg/kg of sugammadex for reversal of pipecuronium-induced neuromuscular blockade
  Interventions: Drug: sugammadex
- placebo group (Placebo Comparator): 3 ml of saline (placebo) for reversal of pipecuronium-induced neuromuscular blockade
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sugammadex — Anesthetised patients will receive a single intubation dose of succinylcholine (1.0 mg/kg) and maintenance bolus dose of pipecuronium (0.08 mg/kg) to maintain the level of neuromuscular blockade at reappearance of T2 Sugammadex in the dose of 4 mg/kg is to be administered as an intravenous bolus dose at the level of neuromuscular blockade of reappearance of T2 (moderate blockade) by means of TOF-Watch SX after the last dose of pipecuronium according to randomization
  Other Names: Bridion
  Arms: sugammadex group
Drug: placebo — Anesthetised patients will receive a single intubation dose of succinylcholine (1.0 mg/kg) and maintenance bolus dose of pipecuronium (0.08 mg/kg) to maintain the level of neuromuscular blockade at reappearance of T2. 3,0 ml of saline (placebo) is to be administered as an intravenous bolus dose at the level of neuromuscular blockade of reappearance of T2 (moderate blockade) by means of TOF-Watch SX after the last dose of pipecuronium according to randomization
  Arms: placebo group

SUMMARY:
Primary objectives:

1. to investigate the efficacy of sugammadex in dose of 4 mg/kg administered at reappearance of T2 for reversal of pipecuronium-induced neuromuscular blockade in subjects undergoing abdominal surgery under general anesthesia
2. to evaluate the safety and tolerability of a single dose of 4 mg/kg sugammadex administered at reappearance of T2 for reversal of pipecuronium-induced neuromuscular blockade

Secondary objectives:

1. to evaluate the time from the start of sugammadex or placebo administration to the time of extubation and to the time of recovery of TOF ratio to ≥ 0.9

Exploratory objectives:

1. to evaluate the Operating Room (OR) and Post Anesthetic Care Unit (PACU) length of stay after the end of surgery in subjects with pipecuronium induced neuromuscular blockade reversed by 4.0 mg.kg-1 sugammadex compared to placebo (saline)
2. compare the number of patients extubated in the OR after the reversal by sugammadex or placebo, evaluate the TOF ratio at the time of extubation

Clinical hypothesis:

1. Sugammadex has to be effective and well tolerated for reversal of pipecuronium-induced blockade

DETAILED DESCRIPTION:
Sugammadex is the first selective relaxant binding agent indicated for reversal of rocuronium and vecuronium-induced blockade.

At the same time sugammadex is able to form the complexes with other aminosteroid-based muscle relaxants including long acting NMBAs* such as pancuronium 1,2.

Still there are only limited data on the efficacy of sugammadex with pancuronium and no data on the efficacy of sugammadex with other aminosteroid-based long acting NMBA - pipecuronium which is still widely used in Russia (as well as in the other former Soviet Union Countries and Eastern Europe countries). In the only study evaluating efficacy of sugammadex with pancuronium has been shown that moderate pancuronium-induced blockade is effectively reversed in less than 3 minutes with a sugammadex dose of 4.0 mg/kg 3. In this respect it would be interesting in this study to evaluate the efficacy of sugammadex with pipecuronium.

It is also very well known that the incidence of postoperative residual blockade (and its complications) is higher when the long acting NMBAs such as pancuronium and pipecuronium are used 4,5,6,7. So the possibility to use sugammadex for reversal of pipecuronium-induced blockade could help to reduce the incidence of residual blockade and related complications.

The effectiveness of sugammadex for the reversal of long acting NMBAs such as pipecuronium at the same time would be significant in light of the limitations of cholinesterase inhibitors. These drugs are more often administered after the long acting NMBAs taking into account their prolonged clinical duration of action.

It is expected that the dose of sugammadex 4 mg/kg will allow to recover the TOF ratio to 0.9 in less than 4 min and in this case this time will be similar to the recovery time after moderate pancuronium-induced blockade.

*NMBAs-neuromuscular blocking agents

2.3 Study Design

1. A single center, randomized, parallel-group, placebo-controlled, safety-assessor (single) blinded trial
2. Adult patients undergoing abdominal surgery under general anesthesia who receive succinylcholine for tracheal intubation and pipecuronium for maintenance of neuromuscular blockade. Planned number of subjects - 42
3. Patients will be randomised into 2 groups to receive at the end of surgery 4 mg/kg of sugammadex or 3 ml of saline (placebo) for reversal of pipecuronium-induced neuromuscular blockade. According to the sample size justification randomization will be done with the ratio of 1:2 - 14 patients will be enrolled in the placebo group and 28 patients - in sugammadex group
4. Neuromuscular function will be monitored using the objective neuromuscular monitoring with the TOF-Watch® SX acceleromyograph at the adductor pollicis muscle, starting after induction of anesthesia (before succinylcholine and pipecuronium administration) and continuing at least until recovery of the TOF ratio to 0.9
5. The primary efficacy variable is the time from the start of sugammadex or placebo administration (reappearance of T2) to recovery of the TOF ratio to 0.9
6. The secondary efficacy variable is the time from the start of sugammadex or placebo administration to the time of extubation
7. Safety assessment is going to be done in order to evaluate the safety and tolerability of sugammadex for reversal of pipecuronium-induced neuromuscular blockade (analysis of AEs and vital signs)

   Safety variables:
   * Vital signs, i.e. heart rate and blood pressure (at screening, pre-pipecuronium, pre-sugammadex or pre-placebo, at 2, 5, 10, and 30 minutes post-sugammadex or post-placebo, and at the post-anesthetic visit)
   * Physical examination (at screening, at the post-anesthetic visit)
   * Pre-treatment (serious) events (from signing informed consent until administration of sugammadex or placebo) and (serious) adverse events ((S)AEs, from administration of sugammadex or placebo up to the end of trial)
8. Descriptive Variables:

   * Time from OR admission (physical placement of subject into the OR) to actual OR discharge
   * Time from start of sugammadex or placebo administration to actual OR discharge
   * Time from tracheal extubation to actual OR or PACU discharge
   * Time from PACU admission to actual PACU discharge
   * Number of patients extubated in the OR in both groups

ELIGIBILITY:
Inclusion Criteria:

* Subjects of ASA class 1-3
* Subjects of age ≥ 18 years
* Subjects undergoing abdominal surgery under general anesthesia who receives succinylcholine for tracheal intubation and pipecuronium for maintenance of neuromuscular blockade
* Subjects who have given written informed consent

Exclusion Criteria:

* Subjects in whom a difficult intubation is expected
* Subjects known or suspected to have neuromuscular disorders affecting NMB
* Subjects known or suspected to have a significant renal dysfunction or a severe hepatic dysfunction
* Subjects known or suspected to have (family) history of malignant hyperthermia
* Subjects known or suspected to have an allergy to opioids, muscle relaxants or other medication used during general anesthesia
* Female subjects who are pregnant
* Female subjects who are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
time from the start of sugammadex or placebo administration (reappearance of T2) to recovery of the TOF ratio to 0.9 | during peri-anesthetic period (after the surgery and until 10 hours after the surgery)
  measurement of time from the start of sugammadex or placebo administration (reappearance of T2) to recovery of the TOF ratio to 0.9

SECONDARY OUTCOMES:
time from the start of sugammadex or placebo administration to the time of extubation | during peri-anesthetic period (after the surgery and until 10 hours after the surgery
  measurement of time from the start of sugammadex or placebo administration to the time of extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Central Clinical Hospital #1 of LLC "Russian Railroad", Moscow, Moscow, Russia